CLINICAL TRIAL: NCT03248804
Title: The Effect of Incorporating Soy Protein Foods in the Colorado Diet for Weight Loss and Maintenance.
Brief Title: Effect of Soy Protein and Colorado Diet on Weight Loss and Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: DuPont Nutrition and Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-1666
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Overweight; Obesity; Weight Loss
Keywords: Obesity; Weight Loss; body composition; dietary protein
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Subjects are assigned either to the soy group or the non-soy group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soy Group (Experimental): Subjects in the soy group were asked to participate in the Colorado Diet program and to consume 3 soy food items per day.
  Interventions: Behavioral: Soy group
- Non-soy Group (Other): Subjects in the non-soy group were asked to participate in the Colorado Diet program and to avoid soy food products.
  Interventions: Behavioral: Non-soy group

INTERVENTIONS:
Behavioral: Soy group
  Arms: Soy Group
Behavioral: Non-soy group
  Arms: Non-soy Group

SUMMARY:
Dietary protein is a key element of most effective weight loss regimens. This study will investigate the effects of consuming soy protein on body composition and cardiometabolic health within the context of an effective weight loss and maintenance program called the Colorado Diet.

DETAILED DESCRIPTION:
This is a randomized study involving 60 study subjects (30 per arm). Investigators plan to enroll 72 subjects (36 per arm) in order to allow for any potential drop outs with the goal of 60 study completers. Investigators will compare the efficacy of inducing weight loss of two treatment arms all based on the Colorado Diet. Subjects will be randomly assigned to one of two study arms and instructed to follow the Colorado Diet by participating in weekly Colorado Diet group classes (State of Slim class). There will be 4 classes of 18 subjects each (two classes for each treatment group). Subjects will be followed in the study for 12 months. Subjects will be randomized into one of two treatment groups as follows:

* Group 1 will participate in a State of Slim group class, receive a State of Slim book (describing the Colorado Diet), and will then purchase food items allowed in the Colorado Diet from the lists of acceptable foods in the State of Slim book.
* Group 2 will participate in a State of Slim class, receive the State of Slim book, and be provided soy protein foods to be consumed as part of the Colorado Diet (subjects will receive up to 3 foods with approximately 20g of soy protein each, per day).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 18 - 55 years
2. BMI between 27-40
3. Weight stable (have not lost or gained more than 10 pounds in the last 3 months)
4. Generally healthy
5. Able to exercise 70 minutes per day at moderate intensity
6. Willing and able to participate in a State of Slim group class for the first 16 weeks of the study and willing to participate in 5 study visits over the 12 month study period.

Exclusion Criteria:

1. Pregnant or trying to become pregnant.
2. Diagnosis of type 1 or type 2 diabetes
3. Individuals following a vegetarian only diet
4. Food allergies (to soy, dairy, wheat/gluten, eggs, or peanuts)
5. Taking medications that could cause weight loss or weight gain or alter plasma lipids (such as steroids, tricyclic antidepressants, chemotherapy, antipsychotics, prescribed or over-the-counter weight loss agents, statins, fibrates, niacin, etc). Oral contraceptives can be used as long as subject agrees to not change use of these during the study. Multivitamins containing niacin can be used as long as subject agrees to not change use of these during the study.
6. Known renal disease
7. hypothyroidism
8. Current alcohol or drug abuse or dependence (Subjects who have quit smoking in the last 6 months will be excluded. Smokers whose smoking habits have been stable for the last 6 months and which remain stable during the study can be included).
9. Any medical condition for which following a diet and/or 70 minutes of exercise daily would be inadvisable
10. LDL cholesterol levels above 190 mg/dl or triglycerides above 400 mg/dl.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2016-10-29 (Actual); Study Completion 2016-10-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in % body weight at the end of a 16 week period | at month 4
Change from baseline in body fat at the end of 16 week period | at month 4
Change from baseline in % body weight at the end of a 52 week period | at month 12
Change from baseline in body fat at the end of a 52 week period | at month 12
Change from baseline in lipid panel results at end of 16 week period (total cholesterol) | at month 4
Change from baseline in lipid panel results at end of 52 week period (total cholesterol) | at month 12
Change from baseline in lipid panel results at end of 16 week period (LDL) | at month 4
Change from baseline in lipid panel results at end of 52 week period (LDLl) | at month 12
Change from baseline in lipid panel results at end of 16 week period (HDL) | at month 4
Change from baseline in lipid panel results at end of 52 week period (HDL) | at month 12
Change from baseline in lipid panel results at end of 16 week period (triglycerides) | at month 4
Change from baseline in lipid panel results at end of 52 week period (triglycerides) | at month 12

CONTACTS AND LOCATIONS:
Overall Officials: James O Hill, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Anschutz Health and Wellness Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
Banked blood samples may be shared with other researchers (with subject consent)

REFERENCES:
- [Background] Anderson GH, Moore SE. Dietary proteins in the regulation of food intake and body weight in humans. J Nutr. 2004 Apr;134(4):974S-9S. doi: 10.1093/jn/134.4.974S. PMID 15051857
- [Background] Anderson GH, Tecimer SN, Shah D, Zafar TA. Protein source, quantity, and time of consumption determine the effect of proteins on short-term food intake in young men. J Nutr. 2004 Nov;134(11):3011-5. doi: 10.1093/jn/134.11.3011. PMID 15514267
- [Background] Anderson JW, Johnstone BM, Cook-Newell ME. Meta-analysis of the effects of soy protein intake on serum lipids. N Engl J Med. 1995 Aug 3;333(5):276-82. doi: 10.1056/NEJM199508033330502. PMID 7596371
- [Background] Anthony TG, McDaniel BJ, Knoll P, Bunpo P, Paul GL, McNurlan MA. Feeding meals containing soy or whey protein after exercise stimulates protein synthesis and translation initiation in the skeletal muscle of male rats. J Nutr. 2007 Feb;137(2):357-62. doi: 10.1093/jn/137.2.357. PMID 17237311
- [Background] Arciero PJ, Baur D, Connelly S, Ormsbee MJ. Timed-daily ingestion of whey protein and exercise training reduces visceral adipose tissue mass and improves insulin resistance: the PRISE study. J Appl Physiol (1985). 2014 Jul 1;117(1):1-10. doi: 10.1152/japplphysiol.00152.2014. Epub 2014 May 15. PMID 24833780
- [Background] Baer DJ, Stote KS, Paul DR, Harris GK, Rumpler WV, Clevidence BA. Whey protein but not soy protein supplementation alters body weight and composition in free-living overweight and obese adults. J Nutr. 2011 Aug;141(8):1489-94. doi: 10.3945/jn.111.139840. Epub 2011 Jun 15. PMID 21677076
- [Background] Barkeling B, Rossner S, Bjorvell H. Effects of a high-protein meal (meat) and a high-carbohydrate meal (vegetarian) on satiety measured by automated computerized monitoring of subsequent food intake, motivation to eat and food preferences. Int J Obes. 1990 Sep;14(9):743-51. PMID 2228407
- [Background] Booth DA, Chase A, Campbell AT. Relative effectiveness of protein in the late stages of appetite suppression in man. Physiol Behav. 1970 Nov;5(11):1299-302. doi: 10.1016/0031-9384(70)90044-2. No abstract available. PMID 5524514
- [Background] Bowen J, Noakes M, Clifton PM. Appetite regulatory hormone responses to various dietary proteins differ by body mass index status despite similar reductions in ad libitum energy intake. J Clin Endocrinol Metab. 2006 Aug;91(8):2913-9. doi: 10.1210/jc.2006-0609. Epub 2006 May 30. PMID 16735482
- [Background] Brown EC, DiSilvestro RA, Babaknia A, Devor ST. Soy versus whey protein bars: effects on exercise training impact on lean body mass and antioxidant status. Nutr J. 2004 Dec 8;3:22. doi: 10.1186/1475-2891-3-22. PMID 15588291
- [Background] Elia D, Stadler K, Horvath V, Jakus J. Effect of soy- and whey protein-isolate supplemented diet on the redox parameters of trained mice. Eur J Nutr. 2006 Aug;45(5):259-66. doi: 10.1007/s00394-006-0593-z. Epub 2006 Mar 30. PMID 16575496
- [Background] Kalman D, Feldman S, Martinez M, Krieger DR, Tallon MJ. Effect of protein source and resistance training on body composition and sex hormones. J Int Soc Sports Nutr. 2007 Jul 23;4:4. doi: 10.1186/1550-2783-4-4. PMID 17908338
- [Background] Latner JD, Schwartz M. The effects of a high-carbohydrate, high-protein or balanced lunch upon later food intake and hunger ratings. Appetite. 1999 Aug;33(1):119-28. doi: 10.1006/appe.1999.0237. PMID 10447984
- [Background] Marmonier C, Chapelot D, Louis-Sylvestre J. Effects of macronutrient content and energy density of snacks consumed in a satiety state on the onset of the next meal. Appetite. 2000 Apr;34(2):161-8. doi: 10.1006/appe.1999.0302. PMID 10744905
- [Background] Paddon-Jones D, Westman E, Mattes RD, Wolfe RR, Astrup A, Westerterp-Plantenga M. Protein, weight management, and satiety. Am J Clin Nutr. 2008 May;87(5):1558S-1561S. doi: 10.1093/ajcn/87.5.1558S. PMID 18469287
- [Background] Tang JE, Moore DR, Kujbida GW, Tarnopolsky MA, Phillips SM. Ingestion of whey hydrolysate, casein, or soy protein isolate: effects on mixed muscle protein synthesis at rest and following resistance exercise in young men. J Appl Physiol (1985). 2009 Sep;107(3):987-92. doi: 10.1152/japplphysiol.00076.2009. Epub 2009 Jul 9. PMID 19589961
- [Background] Porrini M, Santangelo A, Crovetti R, Riso P, Testolin G, Blundell JE. Weight, protein, fat, and timing of preloads affect food intake. Physiol Behav. 1997 Sep;62(3):563-70. doi: 10.1016/s0031-9384(97)00162-5. PMID 9272665
- [Background] Rolls BJ, Hetherington M, Burley VJ. The specificity of satiety: the influence of foods of different macronutrient content on the development of satiety. Physiol Behav. 1988;43(2):145-53. doi: 10.1016/0031-9384(88)90230-2. PMID 3212049
- [Background] Sites CK, Cooper BC, Toth MJ, Gastaldelli A, Arabshahi A, Barnes S. Effect of a daily supplement of soy protein on body composition and insulin secretion in postmenopausal women. Fertil Steril. 2007 Dec;88(6):1609-17. doi: 10.1016/j.fertnstert.2007.01.061. Epub 2007 Apr 6. PMID 17412329
- [Background] Veldhorst MA, Nieuwenhuizen AG, Hochstenbach-Waelen A, van Vught AJ, Westerterp KR, Engelen MP, Brummer RJ, Deutz NE, Westerterp-Plantenga MS. Dose-dependent satiating effect of whey relative to casein or soy. Physiol Behav. 2009 Mar 23;96(4-5):675-82. doi: 10.1016/j.physbeh.2009.01.004. PMID 19385022
- [Background] Westerterp-Plantenga MS, Nieuwenhuizen A, Tome D, Soenen S, Westerterp KR. Dietary protein, weight loss, and weight maintenance. Annu Rev Nutr. 2009;29:21-41. doi: 10.1146/annurev-nutr-080508-141056. PMID 19400750
- [Background] Hill, JH, Blundell, JE. Macronutrients and satiety: The effects of a high-protein or high-carbohydrate meal on subjective motivation to eat and food preferences. Nutr. Behav. 3: 133-144, 1986.
- [Background] Peters, JC. Control of Energy Balance. Biochemical, physiological, molecular aspects of human nutrition 2nd edition, M.H. Stipanuk ed. Saunders Elsevier: 618-639, 2006.
- [Result] Speaker KJ, Sayer RD, Peters JC, Foley HN, Pan Z, Wyatt HR, Flock MR, Mukherjea R, Hill JO. Effects of consuming a high-protein diet with or without soy protein during weight loss and maintenance: a non-inferiority, randomized clinical efficacy trial. Obes Sci Pract. 2018 May 21;4(4):357-366. doi: 10.1002/osp4.278. eCollection 2018 Aug. PMID 30151230